CLINICAL TRIAL: NCT01665872
Title: New Haven Mental Health Outreach for MotherS (MOMS) Partnership
Brief Title: New Haven MOMS Partnership
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Office of Research on Women's Health (ORWH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1010007484; 5CCEWH1110210501 (Other Grant/Funding Number: PHS Public Health Service (ORWH))
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Depression; Stress
Keywords: Mothers; Depression; Stress; Trauma; Public Housing
MeSH Terms: conditions — Depression; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Behavioral Group Therapy (Experimental): 8-session Cognitive-Behavioral intervention based on Munoz et al's Mother Baby Manual, modified to meet the needs of mothers of children of all ages residing in public housing in New Haven, CT. Intervention co-facilitated by mental health clinician and a Community Mental Health Ambassador (peer).
  Interventions: Behavioral: Cognitive-Behavioral Group Therapy
- Standard of care - Cognitive-Behavioral Group Therapy (Active Comparator): 8-session Cognitive-Behavioral intervention based on Munoz et al's Mother Baby Manual, modified to meet the needs of mothers of children of all ages residing in public housing in New Haven, CT. Intervention administered by mental health clinician.
  Interventions: Behavioral: Cognitive-Behavioral Group Therapy

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Group Therapy — CBT Group
  Other Names: CBT Group

SUMMARY:
Phase II of the MOMS Partnership aims to:

1. conduct a needs assessment of the mental health of mothers residing in New Haven, CT;
2. provide on-site group intervention services (randomized by housing community) to improve signs/symptoms of depression/stress/trauma among mothers living onsite.

DETAILED DESCRIPTION:
The purpose of this project is to expand and enhance the New Haven Mental health Outreach for Mothers (MOMs) Coalition beyond pregnancy and depression to include a broader definition of mental illness (depressive, anxiety, and substance use disorders), and a larger target population (low-income, racially and ethnically diverse, pregnant and parenting women) in the City of New Haven. Through this expansion, the Coalition will bring together the community of women, their families and advocates, healthcare providers, policy and agency leaders, and academics, to inform the development and conduct of public health approaches around the mental health of low-income, racially and ethnically diverse, pregnant and parenting women. The specific goals of this Phase I proposal are:

1. To conduct a community-led needs assessment on the mental health of low-income, ethnically and racially diverse pregnant and parenting women in the City of New Haven.
2. To provide randomized intervention services to improve signs/symptoms of depression/stress/trauma among mothers living in public housing in New Haven, CT

ELIGIBILITY:
Inclusion Criteria:

* CES-D score >=16
* Child under the age of 18 (participant must be a mother)
* Resident of public housing authority complex in New Haven, CT or an affiliated Section 8 recipient

Exclusion Criteria:

* Positive for psychosis
* Active suicidal ideation
* Non-English or Spanish speakers
* Unable to provide informed consent
* Unwilling to accept randomization
* Moving within the intervention & follow-up period

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan V Smith, MPH, DrPH, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- See also: Study website — http://www.newhavenmomspartnership.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened throughout the community with a needs assessment during the time frame 05/21/2012 through 06/02/2016.
Period: Screening
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Started (Eligibility based on CES-D score, live in public housing site or receive section 8 or RAP.) | 172 | 172
Completed (All participants completed screening.) | 172 | 172
Not Completed | 0 | 0
Period: Treatment
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Started (Participants who started treatment completed an intake (only a subset of those screened).) | 87 | 67
Completed (Attended at least 2 classes in the 8 class Stress Management course) | 72 | 50
Not Completed | 15 | 17
Period: 6 Month Follow-up
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Started (Those eligible for 6 month follow-up, were class completers (as defined above).) | 72 | 50
Completed (Attended and completed the 6 month follow-up assessment.) | 66 | 49
Not Completed | 6 | 1
Period: 12 Month Follow-up
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Started (Those eligible for 12 month follow-up, were class completers (as defined above).) | 72 | 50
Completed (Attended and completed the 12 month follow-up assessment.) | 58 | 47
Not Completed | 14 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cognitive-Behavioral Group Therapy: Stress Management Class delivered in public housing sites by both a clinician and Community Mental Health Ambassador
- Standard of Care - Cognitive-Behavioral Group Therapy: Stress Management Class delivered in public housing sites by only a clinician
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy | Total
Number analyzed (Participants) | 87 | 67 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 87 | 67 | 154
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (11.0) | 39.2 (11.2) | 38.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 67 | 154
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: White, Non-Hispanic | 3 | 5 | 8
  Race / Ethnicity: Black, Non-Hispanic | 68 | 52 | 120
  Race / Ethnicity: White, Hispanic | 11 | 6 | 17
  Race / Ethnicity: Black, Hispanic | 2 | 3 | 5
  Race / Ethnicity: Other | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 87 | 67 | 154
CES-D total score [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiologic Studies Depression Scale (CES-D) is a screening test for depression and depressive disorder. The total score is a sum which ranges from 0-60. Higher scores indicate the presence of more symptomatology.
  Radloff, L.S. (1977) 'The CES-D scale: A self report depression scale for research in the general population'. Applied Psychological Measurement 1: 385-401.
  units on a scale | 28.2 (9.3) | 30.4 (9.8) | 29.2 (9.6)
Total outpatient mental health or substance abuse visits [Mean (Standard Deviation); unit: visits] — Population: We did not have a response from 3 participants in the Cognitive-Behavioral Group Therapy group
  visits
    number analyzed (Participants) | 84 | 67 | 151
    (all) | 4.5 (16.3) | 2.1 (10.0) | 3.4 (13.9)
Parenting Stress Index Short Form: Parental Distress Percentile [Mean (Standard Deviation); unit: percentile] — Parental Distress is a subscale of Parenting Stress Index Short Form by Richard R. Abidin. This subscale contains 12 questions. The score is the sum of all 12 questions that is then translated to percentiles for normative data (provided by the publisher). This subscale measures distress that the parent is experiencing in their role as a parent as a result of factors related to parenting. High scores indicate more distress.
  Percentiles range from 0-100. Population: This measure was only collected on participants whose youngest child was 7 years or younger.
  percentile
    number analyzed (Participants) | 47 | 34 | 81
    (all) | 82.4 (21.2) | 73.9 (28.5) | 78.9 (24.7)
Parenting Stress Index: Parent-Child Dysfunctional Interaction Percentile [Mean (Standard Deviation); unit: percentile] — Parent-Child Dysfunctional Interaction is a subscale (12 questions) of Parenting Stress Index Short Form by Richard R. Abidin. The score is the sum of all 12 questions. This score is then translated to percentiles for normative data (provided by the publisher). The Parent-Child Dysfunctional Interaction subscale measures the parent's perception that a child does or does not meet their expectations and if interactions with the child are reinforcing to the parent. High scores indicate a parent-child bond that is threatened or not adequately established. Percentiles range from 0-100. Population: This measure was only collected on participants whose youngest child was 7 years or younger.
  percentile
    number analyzed (Participants) | 47 | 34 | 81
    (all) | 61.4 (30.0) | 59.6 (33.3) | 60.7 (31.2)
Parenting Stress Index: Difficult Child Percentile [Mean (Standard Deviation); unit: percentile] — The Difficult Child is a subscale of Parenting Stress Index Short Form by Richard R. Abidin that is created from 12 questions. The score is the sum of all 12 questions. This score is then translated to percentiles for normative data (provided by the publisher). The Difficult Child subscale looks at behavioral characteristics of children (temperament but also patterns of behavior) that make the child easy or difficult to manage. Higher scores generally indicate the parent is experiencing difficulty managing the child's behavior.
  Percentiles range from 0-100. Population: This measure was only collected on participants whose youngest child was 7 years or younger.
  percentile
    number analyzed (Participants) | 47 | 34 | 81
    (all) | 62.0 (33.6) | 58.9 (31.4) | 60.7 (32.5)
Parenting Stress Index Short Form: Total Score Percentile [Mean (Standard Deviation); unit: percentile] — Parenting Stress Index Short Form by Richard R. Abidin, contains a total score which is the sum of all 36 questions. The score is then translated to percentiles for normative data (provided by the publisher). The total score is intended to represent an overall level of parenting stress that the individual is experiencing. A score at or above 90 indicates experiencing clinically significant levels of stress.
  Percentiles range from 0-100. Population: This measure was only collected on participants whose youngest child was 7 years or younger.
  percentile
    number analyzed (Participants) | 47 | 34 | 81
    (all) | 75.8 (27.6) | 71.4 (29.2) | 74.0 (28.2)
Gainful Employment [Count of Participants; unit: Participants] — Do you work 15 hours or more per week for pay?
  Participants
    Yes | 16 | 8 | 24
    No | 71 | 59 | 130

OUTCOME MEASURES:

1. Primary Outcome: Total Outpatient Mental Health or Substance Abuse Visits
Description: Self-report questionnaire which measure attitudes toward seeking mental health treatment. This is defined by looking at total number of outpatient mental health or substance abuse treatment visits in the past year.
Time Frame: 1 year
Population: Participants who attended the 12 month follow-up assessment and completed the questions regarding mental health and substance abuse visits.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Number analyzed (Participants) | 68 | 50
visits | 1.03 (2.95) | 1.21 (6.0)
Statistical Analysis 1: Comparison: Cognitive-Behavioral Group Therapy vs Standard of Care - Cognitive-Behavioral Group Therapy; Test type: Equivalence — A Wilcoxon-Mann-Whitney test was used to test for equivalence. A p-value of 0.05 was used to determine if the difference falls out of the equivalence limits; p = 0.172, t-test, 2 sided

2. Primary Outcome: Depressive and Anxiety Symptoms (CES-D)
Description: The Center for Epidemiologic Studies Depression Scale (CES-D) is a screening test for depression and depressive disorder. The total score is a sum which ranges from 0-60. Higher scores indicate the presence of more symptomatology.
  Radloff, L.S. (1977) 'The CES-D scale: A self report depression scale for research in the general population'. Applied Psychological Measurement 1: 385-401.
Time Frame: approximately 1 year
Population: Participants who attended the 12 month follow-up assessment.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Number analyzed (Participants) | 58 | 47
units on a scale | 13 [9 to 21] | 15 [9 to 24]
Statistical Analysis 1: Comparison: Cognitive-Behavioral Group Therapy vs Standard of Care - Cognitive-Behavioral Group Therapy; Are CES-D scores at 12 months different between groups?; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.5337, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Parenting Stress
Description: Parenting Stress Index Short Form by Richard R. Abidin (total score (36 questions) and 3 subscales (12 questions each) was used to describe parenting stress. Scores were created by summing the responses and then translated to percentiles for normative data (provided by the publisher). The total score represents an overall level of experienced parenting stress. A score 90 or above indicates experiencing clinically significant levels of stress. The subscale Parental Distress measures distress that the parent is experiencing related to parenting. High scores indicate more distress. The Parent-Child Dysfunctional Interaction subscale measures the parent's perception regarding a child meeting expectations and reinforcing interactions with the child. High scores indicate a parent-child bond that is threatened or not adequately established. The Difficult Child subscale looks at behavioral characteristics of children. Higher scores indicating difficulty managing the child's behavior.
Time Frame: 1 year
Population: This questionnaire was only administered to participants who had a child 8 years or older. Results are from participants who attended the 12 month follow-up assessment.
Measure: Median (Inter-Quartile Range); unit: percentile
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Number analyzed (Participants) | 28 | 19
percentile
  Parental Distress | 65 [32.5 to 90] | 50 [1 to 70]
  Parent-Child Dysfunctional Interaction | 42.5 [7.5 to 85] | 20 [5 to 70]
  Difficult Child | 57.5 [15 to 80] | 10 [1 to 75]
  Total | 65 [25 to 85] | 15 [5 to 65]
Statistical Analysis 1: Comparison: Cognitive-Behavioral Group Therapy vs Standard of Care - Cognitive-Behavioral Group Therapy; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0920, Wilcoxon (Mann-Whitney) — This test looks at a difference in Parental Distress at the 12 month follow-up between groups
Statistical Analysis 2: Comparison: Cognitive-Behavioral Group Therapy vs Standard of Care - Cognitive-Behavioral Group Therapy; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.3352, Wilcoxon (Mann-Whitney) — This test looks at a difference in Parent-Child Dysfunctional Interaction at the 12 month follow-up between groups
Statistical Analysis 3: Comparison: Cognitive-Behavioral Group Therapy vs Standard of Care - Cognitive-Behavioral Group Therapy; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0404, Wilcoxon (Mann-Whitney) — This test looks at a difference in Difficult Child at the 12 month follow-up between groups
Statistical Analysis 4: Comparison: Cognitive-Behavioral Group Therapy vs Standard of Care - Cognitive-Behavioral Group Therapy; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0915, Wilcoxon (Mann-Whitney) — This test looks at a difference in PSI total score (percentile) at the 12 month follow-up between groups

4. Primary Outcome: Gainful Employment
Description: Measure of subject's ability to obtain gainful employment
Time Frame: 1 year
Population: Participants who attended 12 month follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Number analyzed (Participants) | 58 | 47
Participants
  Work 15 hours or more for pay | 19 | 11
  Does not work 15 hours or more for pay | 39 | 36
Statistical Analysis 1: Comparison: Cognitive-Behavioral Group Therapy vs Standard of Care - Cognitive-Behavioral Group Therapy; Test type: Equivalence — Chi-square was used with a p-value of 0.05 to determine if the difference was statistically greater than 0; p = 0.2914, Chi-squared

5. Primary Outcome: Implementation Cost
Description: The implementation cost of providing a 8 session Stress Management (SM) Series (with 1 active series at a time) for both Standard of care with only a clinician, and also for a clinician and CMHA. The implementation costs include startup costs and on-going costs. On-going costs include staff salary, travel time, cell phones, space, and materials).
Time Frame: 1 series
Population: Since we are looking at implementation cost this measure isn't participant based, but calculated on what it would cost to run one series.
Measure: Number; unit: American Dollars
Units Other Than Participants: 1 SM series
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
Number analyzed (Participants) | NA | NA
Number analyzed (1 SM series) | 1 | 1
American Dollars | 11350 | 10471

ADVERSE EVENTS:
Time Frame: Adverse event data was monitored for all enrolled participants beginning at enrollment. This continued through engagement in the intervention and all follow-up (1 year post intervention).
Description: The definition does not differ.
  Methods for reporting adverse events: any serious, unanticipated and related adverse events or unanticipated problems involving risks to subjects or others will be reported in writing within 48 hours to the HIC and any appropriate funding and regulatory agencies. Fellow investigators and study personnel will be informed through regular study meetings and study sponsors will be informed within 5 days of the event becoming known to the principal investigator.
Arm/Group | Cognitive-Behavioral Group Therapy | Standard of Care - Cognitive-Behavioral Group Therapy
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/67
Other Adverse Events (participants affected / at risk) | 0/87 | 0/67

LIMITATIONS AND CAVEATS:
Limitations include subjects self-selected to participate and uncertainty in the representativeness of our sample to all residents of public housing. The ICER could not be calculated due to similarity in CES-D scores in both groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No